CLINICAL TRIAL: NCT07266714
Title: Ultrasound-guided vs Conventional Intraarticular Injection of Hyaluronic Acid for Management of Temporomandibular Joint Internal Derangement
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhannad (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Sponsor-Investigator, Muhannad, B.D.S( Aljouf University, 2021. Sakaka, KSA) Master Dgree at Oral surgery department (2022) Affiliation: Mansoura University, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0109024OS
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-09

CONDITIONS: Anterior Disk Displacement TMJ
Keywords: Temporomandibular Joint, Disc displacement with reduction, Ultrasound, Hyaluronic acid.
MeSH Terms: interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided itra-articular injection of hyaluronic acid (Experimental)
  Interventions: Device: Ultrasound guided injection with hyaluronic acid
- Conventional intra-articular injection of hyaluronic acid (Experimental)
  Interventions: Other: Conventional

INTERVENTIONS:
Device: Ultrasound guided injection with hyaluronic acid — Ultrtasound Guided injection of Hyaluronic Acid
  Arms: Ultrasound guided itra-articular injection of hyaluronic acid
Other: Conventional — Conventional injection of hyaluronic Acid
  Arms: Conventional intra-articular injection of hyaluronic acid

SUMMARY:
The aim of the study will be to evaluate the clinical efficacy of using ultrasound guidance during intra-articular injection of hyaluronic acid in the management of patients with TMJ internal derangement.

DETAILED DESCRIPTION:
The temporomandibular joint (TMJ) represents one of the most biomechanically sophisticated and functionally critical articulations in the human body, serving as the primary interface between the mandible and the cranium.

This synovial joint facilitates essential orofacial functions including mastication, phonation, deglutition, and emotional expression through its unique ginglymoarthrodial (hinge-gliding) motion.

Temporomandibular disorders (TMDs) constitute a major public health burden, with epidemiological studies reporting prevalence rates ranging from 5% to 12% in global populations, though subclinical manifestations may affect up to 40% of adults.

The socioeconomic impact is substantial, with chronic TMD patients demonstrating significantly reduced quality-of-life indices comparable to conditions like rheumatoid arthritis, primarily due to persistent pain, functional limitations, and comorbidities with tension-type headaches and sleep disturbances.

Historically, TMJ research evolved from purely mechanical models to contemporary biopsychosocial paradigms that acknowledge multifactorial etiology.

Modern diagnostic frameworks, notably the Diagnostic Criteria for TMD (DC/TMD), emphasize the interplay between articular pathophysiology (e.g., disc displacement, osteoarthritis) and psychosocial dimensions (e.g., catastrophizing, depression), necessitating interdisciplinary management strategies.

Advances in molecular biology have elucidated genetic predispositions (e.g., COMT gene polymorphisms) and inflammatory cascades (IL-1β, TNF-α) that modulate pain sensitization and tissue degeneration.

Concurrently, innovations in diagnostic imaging-particularly dynamic MRI and cone-beam computed tomography (CBCT)-have revolutionized the evaluation of joint kinematics and microarchitecture, enabling earlier detection of degenerative changes.

The clinical management landscape continues to evolve toward minimally invasive biotherapies (e.g., platelet-rich plasma injections) and personalized rehabilitation protocols, though significant challenges persist in predicting treatment responsiveness.

Future research imperatives include validating biomarkers for early TMD detection, optimizing tissue-engineering approaches for condylar regeneration, and integrating artificial intelligence for phenotyping heterogeneous patient subgroups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that will be diagnosed disc displacement confirmed clinically and by Magnetic Resonance Imaging (MRI).
2. Patient not responding to conservative therapy
3. Patients age must be (18 - 50).
4. Patients having painful joint, clicking sound, with or without limited mouth opening.
5. Patient's ability and desire to complete the treatment protocol and follow-up visits.

Exclusion Criteria:

1. Patient with an inflammatory or connective tissue disease
2. Patient with previous invasive TMJ surgical procedure.
3. Patient with Neurologic disorders
4. History of injection of any substance into the target TMJ during previous 6 months.
5. Patient with a history of bony adhesion.
6. Malignant disease in the head and neck region.
7. Patient with a psychological problem.
8. Patients having gross mechanical restrictions and condylar fracture

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Pain (Visual Analogue Scale) | preoperative and postoerative after 1 week, 3 month and 6 month
  Pain intensity will be assessed by visual analog scale (VAS) score. Zero score for no pain and 10 score for worst pain experienced
Clicking sound | preoperative and postoerative after 1 week, 3 month and 6 month
  Clicking sound will be assessed as to its presence = 1 or absence = 0.
Maximum inter-incisal opening (MIO) | preoperative and postoerative after 1 week, 3 month and 6 month
  will be measured by Vernier caliper as the vertical distance in millimeters between the maxillary and mandibular incisal edges of the central incisors.
Range of lateral mandibular excursions | preoperative and postoerative after 1 week, 3 month and 6 month
  will be masseured by Vernier caliper as the horizontal distance in millimeter from maxillary mid line to mandibular mid line with the patient first moving the mandible to one side than to the other at the maximum extend

CONTACTS AND LOCATIONS:
Overall Officials: Sally Elsayed Abdelsameaa, Assistant Professor, Principal Investigator — Mansoura University; Muhammad Adel Al-Hawari, Lecturer, Principal Investigator — Mansoura University; Ayman Ahmed Yaseen, Lecturer, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided